CLINICAL TRIAL: NCT06857942
Title: A Phase 4, Prospective, Open-Label, Single Arm Study to Assess the Effectiveness of Tirzepatide After Initiation of Ixekizumab in Adult Participants With Moderate-to-Severe Plaque Psoriasis and Obesity or Overweight in Clinical Practice
Brief Title: A Study to Investigate the Effectiveness of Tirzepatide (LY3298176) Following Initiation of Ixekizumab (LY2439821) in Participants With Moderate-to-Severe Plaque PsO and Obesity or Overweight in Clinical Practice (TOGETHER AMPLIFY-PsO)
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 27319; I1F-MC-RHDD (Other: Eli Lilly and Company)
Record Dates: First submitted 2025-03-03; First posted 2025-03-05 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Psoriasis; Overweight or Obesity
MeSH Terms: conditions — Psoriasis; Overweight; Obesity | interventions — Tirzepatide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Tirzepatide (Experimental): Participants will continue to receive ixekizumab and take tirzepatide subcutaneously (SC) as per label.
  Interventions: Drug: Tirzepatide

INTERVENTIONS:
Drug: Tirzepatide — Administered SC
  Other Names: LY3298176

SUMMARY:
The main purpose of this study is to assess the effectiveness of adding tirzepatide to ixekizumab therapy in standard clinical practice in participants with moderate-to-severe plaque PsO and obesity or overweight with at least 1 weight-related comorbidity.

The study will last up to 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Have a diagnosis of moderate-to-severe plaque PsO, as defined by a dermatologist or other experienced clinician treated PsO (for example, allergologist, nurse practitioner or physician assistant)
* Have body mass index (BMI) of 30 kilograms per meter squared (kg/m²) or greater (obesity) or 27 kg/m² to <30 kg/m² (overweight) in the presence of at least 1 weight-related comorbid condition (hypertension, dyslipidemia, type 2 diabetes mellitus, obstructive sleep apnea, or cardiovascular diseases).
* Must have initiated treatment with ixekizumab for approximately 3 months (± 1 month) prior to decision to add tirzepatide.
* Must be able to initiate tirzepatide (Day 0) within 30 days of treatment decision (baseline/screening).

Exclusion Criteria:

* Have currently received ixekizumab for more than 4 months or less than 2 months.
* Have had any exposure to tirzepatide or other glucagon-like peptide-1 receptor agonist (GLP-1 RAs), for example, dulaglutide, liraglutide, or semaglutide.
* Are currently enrolled in any other clinical study.

Other exclusions

* Have a known hypersensitivity to tirzepatide or to any of its component.
* Have a personal or family history of medullary thyroid cancer.
* Have multiple endocrine neoplasia type 2.
* Have type I diabetes mellitus.
* Have a history of chronic or acute pancreatitis at any time before screening (Visit 1).
* Have a history of proliferative diabetic retinopathy, diabetic maculopathy, or nonproliferative diabetic retinopathy that requires acute treatment.
* Have a history of ketoacidosis or hyperosmolar state/coma.
* Have a history of severe hypoglycemia and hypoglycemia unawareness within the 6 months before screening.
* Have a history of severe gastrointestinal complications, including gastroparesis, gastroesophageal reflux disease, dyspepsia, chronic nausea/constipation/vomiting.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-03-19 (Actual); Primary Completion 2028-05 (Estimated); Study Completion 2028-05 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants Achieving Dermatology Life Quality Index (DLQI) (0,1) | 12 months
  The DLQI is a simple, patient-reported, 10-item, validated, quality of life questionnaire. Scores range from 0 to 30, with higher scores indicating greater impairment of quality of life.
Percentage of Participants Achieving at least 10% Weight Reduction | 12 months
  Percentage of participants achieving at least 10% weight reduction.

SECONDARY OUTCOMES:
Percentage of Participants Achieving Body Surface Area (BSA) ≤1 % [National Psoriasis Foundation (NPF) treat to target] | Month 6 and Month 12
  The BSA is the arithmetic mean of the affected skin surface based on the assumption that the head represents 10%, upper extremities represent 20%, trunk represents 30%, and lower extremities represent 40% of the total body surface. The BSA is calculated through multiplying the affected BSA in the head, upper extremities, trunk, and lower extremities by the respective total BSA previously indicated and summing together the scores of each body area.
Percentage of Participants Achieving BSA ≤3% (NPF acceptable goal) | Month 6 and Month 12
  The BSA is the arithmetic mean of the affected skin surface based on the assumption that the head represents 10%, upper extremities represent 20%, trunk represents 30%, and lower extremities represent 40% of the total body surface. The BSA is calculated through multiplying the affected BSA in the head, upper extremities, trunk, and lower extremities by the respective total BSA previously indicated and summing together the scores of each body area.
Percentage of Participants Achieving Static Physician's Global Assessment (sPGA) (0,1) | Month 6 and Month 12
  The sPGA is an investigator-administered multi-item scale. It determines the participant's psoriasis (PsO) lesions, overall, at a given time point. Overall lesions are graded for plaque elevation, scaling, and erythema, on a range of clear (0), almost clear (1), mild (2), moderate (3), and severe (4).
Percentage of Participants Achieving DLQI ≤5 | Month 6 and Month 12
  The DLQI is a simple, patient-reported, 10-item, validated, quality of life questionnaire. Scores range from 0 to 30, with higher scores indicating greater impairment of quality of life.
Percentage of Participants Achieving Patient Global Assessment (PatGA) Score ≤2 | Month 6 and Month 12
  The PatGA of Psoriasis is a patient-reported single-item scale. Patient Global Assessments allow for an overall evaluation of disease severity or global impact of the disease from the patient's perspective. Participants are asked to rank the severity of their PsO "today" by selecting a number on a 0-to-5 numeric rating scale, with 0 indicating clear/no PsO and 5 indicating severe PsO.
Mean Percent Change of Weight from Baseline | Baseline, Month 6 and Baseline, Month 12
  Mean percent change of weight from baseline.
Percentage of Participants Achieving DLQI Score (0,1) and Least 10% Weight Reduction | Month 6 and Month 12
  The DLQI is a simple, patient-reported, 10-item, validated, quality of life questionnaire. Scores range from 0 to 30, with higher scores indicating greater impairment of quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 8 AM - 8 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (44):
- United States (43):
  - Medical Dermatology Specialists, Phoenix, Arizona
  - First OC Dermatology Research Inc, Fountain Valley, California
  - Center For Dermatology Clinical Research, Inc., Fremont, California
  - Metropolis Dermatology, Los Angeles, California
  - Northridge Clinical Trials, Northridge, California
  - Alliance for Multispecialty Research, LLC, Fort Myers, Florida
  - NeoClinical Research, Hialeah, Florida
  - Skin Care Research, Hollywood, Florida
  - Encore Medical Research, Hollywood, Florida
  - Palm Harbor Dermatology PA d/b/a TrueBlue Clinical Research, Tampa, Florida
  - TruDerm & TruSpa, Wellington, Florida
  - Southeast Research Specialists, Douglasville, Georgia
  - Dawes Fretzin Clinical Research Group, LLC, Indianapolis, Indiana
  - The Indiana Clinical Trials Center, PC, Plainfield, Indiana
  - Equity Medical - Bowling Green, Bowling Green, Kentucky
  - Dermatology and Skin Cancer Specialists, LLC, Rockville, Maryland
  - Metro Boston Clinical Partners, Brighton, Massachusetts
  - David Fivenson, MD, PLC, Ann Arbor, Michigan
  - Great Lakes Research Group, Inc., Bay City, Michigan
  - The Derm Institute of West Michigan, Caledonia, Michigan
  - Skin Cancer and Dermatology Institute - Reno, Reno, Nevada
  - Stracskin, Portsmouth, New Hampshire
  - Psoriasis Treatment Center of Central New Jersey, East Windsor, New Jersey
  - Care Access - Hoboken, Hoboken, New Jersey
  - Equity Medical, New York, New York
  - Revival Research Institute, LLC, Cary, North Carolina
  - Onsite Clinical Solutions - Huntersville, Huntersville, North Carolina
  - Optima Research - Boardman, Boardman, Ohio
  - Oregon Dermatology and Research Center, Portland, Oregon
  - Dermatology Associates of Plymouth Meeting, Plymouth Meeting, Pennsylvania
  - Columbia Dermatology & Aesthetics, Columbia, South Carolina
  - Alliance for Multispecialty Research, LLC, Myrtle Beach, South Carolina
  - DelRicht Research - Thompson's Station, Smyrna, Tennessee
  - Bellaire Dermatology Associates, Bellaire, Texas
  - Modern Research Associates, PLLC, Dallas, Texas
  - Center for Clinical Studies, Houston, Texas
  - Austin Institute for Clinical Research, Pflugerville, Texas
  - Texas Dermatology and Laser Specialists, San Antonio, Texas
  - Center for Clinical Studies, Webster, Texas
  - Alliance for Multispecialty Research, LLC, Layton, Utah
  - Tanner Clinic, Layton, Utah
  - Bellevue Dermatology Clinic, Bellevue, Washington
  - Dermatology of Seattle, Burien, Washington
- Office of Dr. Alma M. Cruz, Carolina, Puerto Rico

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and EU, whichever is later. Data will be indefinitely available for requesting.
URL: http://vivli.org/

REFERENCES:
- See also: Related Info — https://trials.lilly.com/en-US/trial/580055